CLINICAL TRIAL: NCT01491984
Title: Effectiveness and Safety of the Levitan FPS Scope for Laryngoscopy and Tracheal Intubation With a Simulated Difficult Airway in Surgical Subjects Under General Anesthesia
Brief Title: Effectiveness and Safety of the Levitan Scope for Laryngoscopy and Tracheal Intubation With a Simulated Difficult Airway
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Ronald George, Primary Investigator, MD, FRCPC, Assistant Professor, IWK Health Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IWK-4668-2009; IWK REB 4668 (Other: IWK REB number)
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Results first posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-02

CONDITIONS: Airway Complication of Anaesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laryngoscopy order: 1) MAC, 2) Levitan (Experimental): Levitan FPS Intubation
  Interventions: Device: Laryngoscopy order: 1) MAC, 2) Levitan; Device: Laryngoscopy order: 1) Levitan, 2) MAC
- Laryngoscopy order: 1) Levitan, 2) MAC (Experimental): Macintosh Intubation
  Interventions: Device: Laryngoscopy order: 1) MAC, 2) Levitan; Device: Laryngoscopy order: 1) Levitan, 2) MAC

INTERVENTIONS:
Device: Laryngoscopy order: 1) MAC, 2) Levitan — Laryngoscopy with MAC, then Levitan
Device: Laryngoscopy order: 1) Levitan, 2) MAC — Laryngoscopy with Levitan, then MAC

SUMMARY:
A laryngoscope is a medical instrument that is used to get a view of the voice box and the space in between the vocal cords. A laryngoscope is used to place a breathing tube into the trachea (windpipe or airway) to protect the patient's airway and provide a way to help a person breathe during surgery; this is called intubation.

DETAILED DESCRIPTION:
A laryngoscope is a medical instrument that is used to get a view of the voice box and the space in between the vocal cords. A laryngoscope is used to place a breathing tube into the trachea (windpipe or airway) to protect the patient's airway and provide a way to help a person breathe during surgery; this is called intubation. The placement of a breathing tube into the windpipe is a skill that is not easily mastered. In fact, the placement is difficult or impossible using the usual technique in 1-3 of every 100 patients. The ease of placing this breathing tube depends in part on how easily and how much of the vocal cords are able to be seen directly using a laryngoscope.

In a small number of patients, the Levitan First Pass Success (FPS) Scope has been shown to be more effective and easier to insert even in patients who have difficult airways. This study will evaluate the use of the LFS compared to the other conventional laryngoscope in subjects with a simulated difficult airway. The goal of this study is to determine the effectiveness and safety of the LFS in a large number of patients with simulated airway difficulties.

The results obtained during the study may provide useful information to health care providers who cannot place a breathing tube in patients that are either in operating rooms or in emergency situations requiring intubation by paramedics. An example would be a trauma situation where a paramedic is having difficulty attempting an intubation when a patients c-spine is being protected from any movements.

The LFS is an affordable and transportable device, which makes this an attractive asset for health providers in smaller community settings or in paramedic vehicles which may not have the capacity to stock or ability to afford a variety of different scopes and must choose a more limited selection.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status I or II (healthy or mild systemic disease, ex. asthma, high blood pressure)
2. Elective surgery requiring endotracheal intubation
3. English speaking
4. Age 16 - 75 years

Exclusion Criteria:

1. Significant gastroesophageal reflux disease (GERD) that may require alternate induction/intubation techniques
2. Prior history of a difficult intubation requiring an awake tracheal intubation
3. Clinical predictors of a potentially difficult intubation requiring an awake intubation
4. BMI > 45 kg/m2 (Obesity is a common and important risk factor for difficult intubation)

Ages: 16 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B George, MD, Principal Investigator — IWK Health Centre

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 29,2009 to March 12, 2010 we recruited women aged 16-75 yrs old, ASA class I-II, and undergoing elective gynecologic surgery at the IWK Health Centre under general anesthesia with planned orotracheal intubation.
Pre-assignment Details: 105 participants were consented and randomized, and of those 11 were withdrawn for either anticipated difficult airway, decreased SpO2, or unavailable staff/equipment. A total of 94 participants started the study protocol. 3 were withdrawn. 91 participants completed the study protocol.
Groups:
- Levitan FPS/Mac Laryngoscope Intubation Order: Intubation with Levitan
  laryngoscopy view with Levitan :
- Macintosh/Levitan FPS Laryngoscope Intubation Order: traditional MAC intubation
  laryngoscopy view with MAC :
Period: Overall Study
Arm/Group | Levitan FPS/Mac Laryngoscope Intubation Order | Macintosh/Levitan FPS Laryngoscope Intubation Order
Started | 49 | 45
Completed | 47 | 44
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intubation Order Levitan/MAC: The LFS is used to guide and confirm endotracheal placement of endotracheal tubes during routine laryngoscopy.
- Intubation Order MAC/Levitan: A size 7.0-mm endotracheal tube with a malleable stylet was used to facilitate Macintosh intubation (standard practice).
- Total: Total of all reporting groups
Arm/Group | Intubation Order Levitan/MAC | Intubation Order MAC/Levitan | Total
Number analyzed (Participants) | 49 | 45 | 94
Age, Customized [Mean (Standard Deviation); unit: years] | 45 (13) | 45 (13) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 45 | 94
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cormack-Lehane Grade
Description: The anesthesiologist graded the laryngeal view after induction of anesthesia using Cormack-Lehane Scale.
  Grade 1 = full view of glottis Grade 2a = partial view of glottis Grade 2b = Only posterior extremity of glottis seen or only arytenoid cartilages Grade 3 = Only epiglottis seen, none of glottis seen Grade 4 = Neither glottis nor epiglottis seen
Time Frame: intraoperative
Measure: Number; unit: participants
Groups:
- Levitan/MAC Intubation: Laryngoscopy with Levitan, then MAC
- MAC/Levitan Intubation: Laryngoscopy with MAC then Levitan
Arm/Group | Levitan/MAC Intubation | MAC/Levitan Intubation
Number analyzed (Participants) | 91 | 94
participants
  Good Laryngoscopic View-Cormack-Lehane grade 1 & 2 | 58 | 53
  Poor Laryngoscopic View-Cormack-Lehane grade 3 & 4 | 33 | 41

2. Secondary Outcome: Number of Intubation Attempts
Description: Number of intubation attempts was recorded after intubation was completed.
Time Frame: intraoperative
Reporting Status: Not Posted

3. Secondary Outcome: Operator Rating of Difficulty
Description: The attending anesthesiologist rated the difficulty in using each technique to intubate the larynx using an 11-point numeric rating scale and a 4-point visual rating scale.
Time Frame: intraoperative
Reporting Status: Not Posted

4. Secondary Outcome: Time to Successful Intubation
Description: Time to successful intubation was documented during the second laryngoscopy and defined as the time from the insertion of the Macintosh laryngoscope into the oral cavity to its removal.
Time Frame: intraoperative
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Levitan FPS Intubation: The LFS is used to guide and confirm endotracheal placement of endotracheal tubes during routine laryngoscopy.
- Macintosh Intubation: A size 7.0-mm endotracheal tube with a malleable stylet was used to facilitate Macintosh intubation (standard practice)
Arm/Group | Levitan FPS Intubation | Macintosh Intubation
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/94
Other Adverse Events (participants affected / at risk) | 0/91 | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No